CLINICAL TRIAL: NCT03554265
Title: Brain and Gut Plasticity in Mild TBI or Post-acute COVID Syndrome Following Growth Hormone Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0313
Record Dates: First submitted 2018-04-09; First posted 2018-06-13 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Traumatic Brain Injury; Fatigue; Cognitive Impairment; COVID-19
Keywords: growth hormone; Traumatic Brain injury; concussion; mTBI; fatigue; cognitive impairment; BIAFAC; COVID-19; post-COVID syndrome; long hauler COVID-19; post-acute sequelae of SARS-CoV-2
MeSH Terms: conditions — Brain Injuries, Traumatic; Fatigue; Cognitive Dysfunction; COVID-19; Brain Concussion | interventions — Human Growth Hormone

STUDY DESIGN:
Intervention Model Description: mTBI patients will be in the growth hormone arm PASC patients will be in the growth hormone arm Control subjects will be in the control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- mTBI subjects (Experimental): mTBI subjects will receive recombinant human growth hormone replacement therapy daily for 6 months.
  Drug: recombinant human growth hormone (rhgH); somatropin, Genotropin
  Dose: month 0 - month 1 will be dosed at 0.4 mg / day month 1 - month 6 will be dosed at 0.6 mg / day
  Interventions: Drug: Somatropin
- Household Control Subjects (No Intervention): household control subjects will not receive any intervention.
- PASC subjects (Experimental): PASC subjects will receive recombinant human growth hormone replacement therapy daily for 9 months.
  Drug: recombinant human growth hormone (rhgH); somatropin, Genotropin
  Dose: month 0 - month 1 will be dosed at 0.4 mg / day month 1 - month 9 will be dosed at 0.6 mg / day
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Genotropin given by injection
  Other Names: Genotropin
  Arms: PASC subjects; mTBI subjects

SUMMARY:
Patients with a history of mild traumatic brain injury (mTBI) or post acute sequelae of SARS-CoV-2 (PASC) and abnormal growth hormone secretion, as measured by glucagon stimulation test, will be treated with replacement growth hormone therapy for a period of 6 months (mTBI) or 9 months (PASC). Testing of cognition, exercise, fatigue, brain activation and morphology, body composition and measurements of quality of life will be performed before and after the treatment period. Fecal sampling for characterization of the GI microbiome will occur monthly over the treatment period. Control subjects will be enrolled and will provide fecal samples monthly for 6 months. GI microbiomes will be compared between mTBI patients, PASC patients and controls at baseline as well as over the treatment period.

DETAILED DESCRIPTION:
The investigators will study subjects (aged 18-70 years) with a history of mild TBI (n=25), post-acute sequelae of SARS-CoV-2 (PASC) (n=25)and healthy controls (n=25). mTBI subjects will undergo a 6-month intervention of rhGH therapy. PASC subjects will undergo a 9-month intervention of rhGH therapy. Controls will be asked to participate in questionnaires, blood draws (amino acid analysis), and fecal sampling (GI microbiome analysis). Controls will not receive any growth hormone treatment.

mTBI group

All patients presenting with a prior mTBI will undergo a phone pre-screen including the Brief Fatigue Inventory (BFI) questions 1-3. If they score ≥ 3 on any BFI questions 1-3, and are interested in participating in the study, they will be scheduled for a formal consenting and medical screening at the UTMB Clinical Research Center (CRC). During the medical screening, eligibility will be confirmed and a glucagon stimulation test (GST) will be performed. A glucagon stimulation with a growth hormone peak of <10 ng/mL is required to qualify for enrollment.

PASC group

All patients presenting with PASC will undergo a phone pre-screen including the Brief Fatigue Inventory (BFI) questions 1-3. If they score ≥ 3 on any BFI questions 1-3, and are interested in participating in the study, they will be scheduled for a formal consenting and medical screening at the UTMB Clinical Research Center (CRC). During the medical screening, eligibility will be confirmed and a glucagon stimulation test (GST) will be performed. A glucagon stimulation with a growth hormone peak of <10 ng/mL is required to qualify for enrollment.

Control group

All controls will undergo a phone pre-screen and if interested in participating in the study, will be scheduled for a formal consenting and medical screening at the UTMB Clinical Research Center (CRC).

Experimental Protocol.

mTBI Group

Before and at completion (month 6) of the rhGH intervention, mTBI subjects will report to the UTMB Institute for Translational Sciences (ITS) Clinical Research Center (CRC) for testing, which will consist of cognitive function assessment (MoCA), determination of brain morphology and connectivity using fMRI, determination of lean mass and fat mass using DEXA, resting energy expenditure, functional testing including leg strength and 6 minute walk test, fatigue measurements, and questionnaires of mood and quality of life, gastrointestinal health, sleep, and food preferences. Blood sampling for measurement of amino acid levels, hormones, and metabolites will be drawn before and 90 minutes (+/- 10 minutes) after a standardized meal. In addition, fecal samples for analysis of the GI microbiome will be collected monthly for the duration of the study. Insulin Growth Factor 1 (IGF-1) levels will monitored at a month 1 safety visit for all mTBI subjects. The month 1 safety visit will occur +/- 5 days from the expected date based on the baseline study visit. The monthly fecal sampling will occur +/- 7 days from the expected date based on the baseline study visit. The month 6 post study will occur +/- 7 days from the expected date based on the baseline study visit. A member of the study team will contact the subject each month to coordinate fecal sample transport to UTMB, check for adverse events and overall well-being, and ensure compliance and ongoing consent.

PASC Group

Before and at month 6 of the rhGH intervention, PASC subjects will report to the UTMB Institute for Translational Sciences (ITS) Clinical Research Center (CRC) for testing, which will consist of cognitive function assessment (MoCA), determination of lean mass and fat mass using DEXA, resting energy expenditure, functional testing including leg strength and 6 minute walk test, fatigue measurements, and questionnaires of mood and quality of life, gastrointestinal health, sleep, and food preferences. Blood sampling for measurement of amino acid levels, hormones, and metabolites will be drawn before and 90 minutes (+/- 10 minutes) after a standardized meal. In addition, fecal samples for analysis of the GI microbiome will be collected monthly for the duration of the study. Insulin Growth Factor 1 (IGF-1) levels will monitored at a month 1 safety visit for all mTBI subjects. The month 1 safety visit will occur +/- 5 days from the expected date based on the baseline study visit. The monthly fecal sampling will occur +/- 7 days from the expected date based on the baseline study visit. The month 6 post study will occur +/- 7 days from the expected date based on the baseline study visit. PASC subjects will continue on rhGH treatment for an additional 3 months. GI microbiome sampling and questionnaires will occur at month 9 and month 12. PASC subjects will have an repeat glucagon stimulation test (GST) to determine growth hormone status at month 12. A member of the study team will contact the subject each month to coordinate fecal sample transport to UTMB, check for adverse events and overall well-being, and ensure compliance and ongoing consent.

Control group

Before and at month 6, controls will report to the UTMB Institute for Translational Sciences (ITS) Clinical Research Center (CRC) for testing, which will consist of questionnaires of food preferences and gastrointestinal health and blood sampling for measurement of amino acid levels, hormones, and metabolites which will be drawn before and 90 minutes (+/ 10 minutes) after a standardized meal. In addition, fecal samples for the analysis of the GI microbiome will be collected monthly for the duration of the study, as well as questionnaire assessing gastrointestinal health. The monthly fecal sampling will occur +/- 7 days from the expected date based on the baseline study visit. The post study (month 6) will occur +/- 7 days from the expected date based on the baseline study visit. A member of the study team will contact the subject each month to coordinate fecal sample transport to UTMB, check for adverse events and overall well-being, and ensure compliance and ongoing consent.

ELIGIBILITY:
mTBI Inclusion criteria

1. Male or female with a diagnosis of mild TBI.
2. At least 6-month post-injury.
3. Ages 18 to 70 years.
4. Participant is willing and able to give informed consent for participation in the study.

mTBI Exclusion criteria

1. Unable to walk unassisted.
2. Significant heart, liver, kidney, blood or respiratory disease.
3. History of chest pain or coronary heart disease.
4. Uncontrolled Diabetes mellitus.
5. Any history of a recently (12 months) diagnosed cancer other than a skin cancer (excluding melanoma).
6. Recent (within 6 months) treatment with anabolic steroids or corticosteroids.
7. Current alcohol or drug abuse.
8. Premorbid history of psychiatric disorder.
9. Premorbid history of head trauma.
10. Pregnancy or become pregnant during the trial.
11. Coumadin because of the risk of bleeding with daily injections of rhGH.
12. Subjects who are deficient in cortisol or thyroid at screening will be excluded until hormone abnormalities have been corrected.
13. Subjects with chronic pain who are being managed with narcotics will be excluded as the effects of central nervous system depressants may interfere with study test results.
14. Subjects with a history of inflammatory bowel disease, Celiac disease or active diverticular disease.
15. Other medical condition or medication administration deemed exclusionary by the study investigators.

Control Inclusion criteria

1. Ages 18 to 70 years.
2. Participant is willing and able to give informed consent for participation in the study.

Control Exclusion criteria

1. Significant heart, liver, kidney, blood or respiratory disease.
2. Uncontrolled Diabetes mellitus.
3. Any history of a recently (12 months) diagnosed cancer other than a skin cancer (excluding melanoma).
4. Recent (within 6 months) treatment with anabolic steroids or corticosteroids.
5. Current alcohol or drug abuse.
6. Premorbid history of psychiatric disorder.
7. Premorbid history of head trauma.
8. Pregnancy or become pregnant during the trial.
9. Subjects who are deficient in thyroid at screening will be excluded until thyroid hormone is replaced.
10. Subjects with a history of inflammatory bowel disease, Celiac disease or active diverticular disease.
11. Other medical condition or medication administration deemed exclusionary by the study investigators.

PASC Inclusion criteria

1. Male or female with a history of COVID with diagnosis confirmed by PCR test.
2. Minimum of 6 months since diagnosis of COVID by PCR test.
3. Ages 18 to 70 years.
4. Score of 3 or higher on any question 1-3 of the Brief Fatigue Inventory (BFI) questionnaire.
5. Participant is willing and able to give informed consent for participation in the study.

PASC Exclusion criteria

1. Current COVID infection.
2. Unable to walk unassisted.
3. Significant heart, liver, kidney, blood or respiratory disease as determined by Principal Investigator.
4. Uncontrolled diabetes mellitus.
5. Any history of a recently (12 months) diagnosed cancer other than a skin cancer (excluding melanoma).
6. Current alcohol or drug abuse.
7. History of psychosis.
8. Pregnancy or become pregnant during the trial.
9. Subjects who are being managed with narcotics will be excluded as the effects of central nervous system depressants may interfere with study test results.
10. Other medical condition or medication administration deemed exclusionary by the study investigators.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Urban, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wright TJ, Sheffield-Moore M, Pyles RB, Randolph KM, McGovern KA, Danesi CP, Lindsay SE, Zaidan MF, Masel BE, Urban RJ. Growth hormone treatment for neurologic symptoms of post-acute sequelae of COVID-19. Clin Transl Sci. 2024 Jun;17(6):e13826. doi: 10.1111/cts.13826. PMID 38894576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for mTBI and community control subjects began August 2018 and ended August 2022.
  Recruitment for PASC subjects began May 2021 and ended September 2022.
Groups:
- mTBI Subjects: mTBI subjects will receive recombinant human growth hormone replacement therapy daily for 6 months.
  Drug: recombinant human growth hormone (rhgH); somatropin, Genotropin
  Dose: month 0 - month 1 will be dosed at 0.4 mg / day month 1 - month 6 will be dosed at 0.6 mg / day
  Somatropin: Genotropin given by injection
- Community Control Subjects: Community control subjects will not receive any intervention.
- PASC Subjects: PASC subjects will receive recombinant human growth hormone replacement therapy daily for 9 months.
  Drug: recombinant human growth hormone (rhgH); somatropin, Genotropin
  Dose: month 0 - month 1 will be dosed at 0.4 mg / day month 1 - month 9 will be dosed at 0.6 mg / day
  Somatropin: Genotropin given by injection
Period: Overall Study
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Started | 28 | 27 | 17
Completed | 26 | 25 | 13
Not Completed | 2 | 2 | 4
Not completed — Withdrawal by Subject | 2 | 2 | 3
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects | Total
Number analyzed (Participants) | 28 | 27 | 17 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 26 | 17 | 70
  >=65 years | 1 | 1 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (12.2) | 43.3 (13.9) | 49.2 (12.1) | 46.7 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 13 | 47
  Male | 11 | 10 | 4 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 28 | 27 | 17 | 72
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 17 | 72
BMI [Mean (Standard Deviation); unit: (kg/m2)] | 28.9 (6.1) | 26.5 (4.0) | 32.0 (7.0) | 28.7 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Lean Body Mass as Measured by Dual Energy X-Ray Absorptiometry (DEXA) at Baseline
Description: Lean body mass will be measured in mTBI and PASC subjects by GE Lunar iDEXA at baseline.
Time Frame: baseline
Population: Community Control subjects did not undergo this procedure.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
kilograms | 49.9 (11.8) |  | 49.6 (13.2)

2. Primary Outcome: Lean Body Mass as Measured by Dual Energy X-Ra Absorptiometry (DEXA) at 6 Months
Description: Lean body mass will be measured in mTBI and PASC subjects by GE Lunar iDEXA after 6 months of growth hormone treatment.
Time Frame: 6 months
Population: Community control subjects did not undergo this procedure.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 25 | 0 | 14
kilograms | 52.3 (11.6) |  | 48.2 (13.2)

3. Primary Outcome: Fat Mass as Measured by Dual Energy X-Ra Absorptiometry (DEXA) at Baseline
Description: Fat mass will be measured in mTBI and PASC subjects by GE Lunar iDEXA at baseline.
Time Frame: baseline
Population: Community controls did not undergo this procedure.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
kilograms | 30.8 (12.5) |  | 38.1 (13.9)

4. Primary Outcome: Fat Mass as Measured by Dual Energy X-Ra Absorptiometry (DEXA) at 6 Months
Description: Fat mass will be measured in mTBI and PASC subjects by GE Lunar iDEXA after 6 months of growth hormone treatment.
Time Frame: 6 months
Population: Community Controls did not undergo this procedure.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 25 | 0 | 14
kilograms | 31.0 (13.3) |  | 34.3 (12.3)

5. Secondary Outcome: Basal Metabolic Rate as Measured by Resting Energy Expenditure at Baseline
Description: Resting Energy Expenditure will be measured by capturing the expired breath of mTBI and PASC subjects while at rest with a metabolic cart over a 30 minute time period. Data will be reported as kilocalories/day.
Time Frame: baseline
Population: Community Control subjects did not undergo this procedure.
Measure: Mean (Standard Deviation); unit: kilocalories per day
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
kilocalories per day | 1484 (260) |  | 1512 (378)

6. Secondary Outcome: Basal Metabolic Rate as Measured by Resting Energy Expenditure at 6 Months
Description: Resting Energy Expenditure will be measured by capturing the expired breath of mTBI and PASC subjects while at rest with a metabolic cart over a 30 minute time period. Data will be reported as kilocalories/day. This will be measured after 6 months of growth hormone treatment in mTBI and PASC subjects only.
Time Frame: 6 months
Population: Community Control subjects did not undergo this procedure. 2 PASC subjects did not undergo 6m measurement due to equipment failure.
Measure: Mean (Standard Deviation); unit: kilocalories per day
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 25 | 0 | 12
kilocalories per day | 1656 (243) |  | 1455 (292)

7. Other Pre Specified Outcome: Cognitive Function as Measured by Montreal Cognitive Assessment at Baseline
Description: The Montreal Cognitive Assessment (MoCA) will be used to assess cognition at baseline in mTBI and PASC subjects only.
  The Montreal Cognitive Assessment (MoCA) is a rapid assessment of cognition. The MoCA consists of 9 questions with the following subcategories: visuospatial/executive, naming, memory, language, abstraction, delayed recall and orientation. The MoCA has been used extensively to detect cognitive impairment in many conditions, including head trauma. Version 7.1 will be used at the Month 0 testing and Version 7.2 will be used at the Month 6 testing. Scores range from 0 to 30, higher score being a better outcome.
Time Frame: baseline
Population: Community control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
score on a scale | 26.0 (2.6) |  | 26.2 (2.9)

8. Other Pre Specified Outcome: Cognitive Function as Measured by Montreal Cognitive Assessment at 6 Months
Description: The Montreal Cognitive Assessment (MoCA) will be used to assess cognition after 6 months of growth hormone treatment in mTBI and PASC subjects only.
  The Montreal Cognitive Assessment (MoCA) is a rapid assessment of cognition. The MoCA consists of 9 questions with the following subcategories: visuospatial/executive, naming, memory, language, abstraction, delayed recall and orientation. The MoCA has been used extensively to detect cognitive impairment in many conditions, including head trauma. Version 7.1 will be used at the Month 0 testing and Version 7.2 will be used at the Month 6 testing. Scores range from 0 to 30, higher score being a better outcome.
Time Frame: 6 months
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 25 | 0 | 14
score on a scale | 26.5 (2.2) |  | 27 (2.3)

9. Other Pre Specified Outcome: Global Fatigue Score as Measured by Brief Fatigue Inventory (BFI) at Baseline
Description: The Brief Fatigue Inventory is a 9 item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life), with "0" being no fatigue and "10" being as bad as you can imagine. The Global Fatigue score is calculated by averaging the answers of all the questions. Brief Fatigue Inventory is measured in mTBI and PASC subjects at baseline.
Time Frame: baseline
Population: Community Controls did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
score on a scale | 6.1 (2.1) |  | 5.7 (2.2)

10. Other Pre Specified Outcome: Global Fatigue Score as Measured by Brief Fatigue Inventory (BFI) at 6 Months
Description: The Brief Fatigue Inventory is a 9 item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life), with "0" being no fatigue and "10" being as bad as you can imagine. The Global Fatigue score is calculated by averaging the answers of all the questions. Brief Fatigue Inventory is measured in mTBI and PASC subjects after 6 months of growth hormone treatment.
Time Frame: 6 months
Population: Community Controls did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 26 | 0 | 14
score on a scale | 3.4 (2.9) |  | 3.4 (2.8)

11. Other Pre Specified Outcome: Global Fatigue Score as Measured by Brief Fatigue Inventory (BFI) at 9 Months
Description: The Brief Fatigue Inventory is a 9 item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life), with "0" being no fatigue and "10" being as bad as you can imagine. The Global Fatigue score is calculated by averaging the answers of all the questions. Brief Fatigue Inventory is measured in PASC subjects after 9 months of growth hormone treatment.
Time Frame: 9 months
Population: Community control subjects did not complete this measure. mTBI subjects did not complete 9m measurements.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 12
score on a scale |  |  | 3.1 (1.9)

12. Other Pre Specified Outcome: Global Fatigue Score as Measured by Brief Fatigue Inventory (BFI) at 12 Months
Description: The Brief Fatigue Inventory is a 9 item questionnaire that assesses perceptual fatigue as well as fatigue interferences (e.g. interference with enjoyment of life), with "0" being no fatigue and "10" being as bad as you can imagine. The Global Fatigue score is calculated by averaging the answers of all the questions. Brief Fatigue Inventory is measured in PASC subjects after 9 months of growth hormone treatment and 3 months off treatment (total time: 12 months).
Time Frame: 12 months
Population: Community control subjects did not complete this measure. mTBI subjects did not complete 12m measurements.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 4.3 (3.0)

13. Other Pre Specified Outcome: Personal Perception of Fatigue as Measured by Multidimensional Fatigue Symptom Inventory - Short Form at Baseline
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
  The MFSI is measured at baseline.
Time Frame: baseline
Population: Community control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
score on a scale | 47.7 (20.1) |  | 44.5 (22.3)

14. Other Pre Specified Outcome: Personal Perception of Fatigue as Measured by Multidimensional Fatigue Symptom Inventory - Short Form at 6 Months
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
  The MFSI is measured after 6 months of growth hormone treatment.
Time Frame: 6 months
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 26 | 0 | 14
score on a scale | 17.7 (27.9) |  | 17.8 (23.9)

15. Other Pre Specified Outcome: Personal Perception of Fatigue as Measured by Multidimensional Fatigue Symptom Inventory - Short Form at 9 Months
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
  The MFSI is measured after 9 months of growth hormone treatment in PASC subjects only.
Time Frame: 9 months
Population: mTBI and community control subjects are complete at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 11.1 (19.6)

16. Other Pre Specified Outcome: Personal Perception of Fatigue as Measured by Multidimensional Fatigue Symptom Inventory - Short Form at 12 Months
Description: Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF) from the Moffitt Cancer Center, University of South Florida The MFSI-SF is a 30 question assessment designed to assess the principal manifestations of fatigue.
  There 5 subscales used to calculate a total score. The subscales are: General Fatigue, Physical Fatigue, Emotional Fatigue, Mental Fatigue, and Vigor (an estimate of the patient's energy level). The total score is calculated with the equation: (general + physical + emotional + mental) - vigor = total score.
  The range of the total score is -24 to 96, with the higher the number meaning more fatigue.
  The MFSI is measured after 9 months of growth hormone treatment and then 3 months without treatment (total 12 months) in PASC subjects only.
Time Frame: 12 months
Population: mTBI and community control subjects are complete at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 21.3 (23.9)

17. Other Pre Specified Outcome: Gastrointestinal Health as Measured by the Gastrointestinal Symptom Rating Scale at Baseline
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The average of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 1 (best outcome) to 75 (worst outcome). GSRS will be measured monthly at baseline mTBI, PASC and control subjects.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 26 | 17
score on a scale | 2.3 (0.72) | 1.51 (0.49) | 2.4 (0.78)

18. Other Pre Specified Outcome: Gastrointestinal Health Measured by the Gastrointestinal Symptom Rating Scale at 6 Months
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The average of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 1 (best outcome) to 7 (worst outcome). GSRS will be measured monthly in all subjects.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 27 | 23 | 14
score on a scale | 1.7 (0.75) | 1.5 (0.55) | 1.8 (0.7)

19. Other Pre Specified Outcome: Gastrointestinal Health Measured by the Gastrointestinal Symptom Rating Scale at 9 Months
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The average of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 1 (best outcome) to 7 (worst outcome). GSRS will be measured in month 9 in PASC subjects only.
Time Frame: 9 months
Population: mTBI and community control subjects complete the study at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 11
score on a scale |  |  | 2.0 (0.99)

20. Other Pre Specified Outcome: Gastrointestinal Health Measured by the Gastrointestinal Symptom Rating Scale at 12 Months
Description: The Gastrointestinal Symptom Rating Scale (GSRS) is a specific 15-item questionnaire. Subjects are asked to numerically score their subjective symptoms on a scale of 1-7 (1 = no discomfort at all; 7 = very severe discomfort) . The average of the scores for all 15 items is regarded as the GSRS total score. Total scores range from 1 (best outcome) to 7 (worst outcome). GSRS will be measured in month 12 in PASC subjects only.
Time Frame: 12 months
Population: mTBI and community control subjects complete the study at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 1.94 (1.2)

21. Other Pre Specified Outcome: Mood Measured by Profile of Mood States at Baseline
Description: Profile of Mood States (POMS) is a questionnaire by MultiHealth Systems, that measures mood. In this 65 item questionnaire, subjects are asked to rate their feelings toward a statement from 0-4, with 0 being "not at all' and 4 being "extremely". There are 6 subscales which include, tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. To calculate the total mood disturbance, which is what is reported here, the subscales tension-anxiety, depression, anger-hostility, fatigue and confusion are summed and vigor is subtracted. The scale range for total mood disturbance is 200 (worst) to -32 (best). POMS will be measured at baseline in mTBI and PASC subjects only.
Time Frame: baseline
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
score on a scale | 49.8 (36.3) |  | 49.6 (45.1)

22. Other Pre Specified Outcome: Mood Measured by Profile of Mood States at 6 Months
Description: Profile of Mood States (POMS) is a questionnaire by MultiHealth Systems, that measures mood. In this 65 item questionnaire, subjects are asked to rate their feelings toward a statement from 0-4, with 0 being "not at all' and 4 being "extremely". There are 6 subscales which include, tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. To calculate the total mood disturbance, which is what is reported here, the subscales tension-anxiety, depression, anger-hostility, fatigue and confusion are summed and vigor is subtracted. The scale range for total mood disturbance is 200 (worst) to -32 (best). POMS will be measured after 6 months of treatment with Growth hormone in mTBI and PASC subjects only.
Time Frame: 6 months
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 25 | 0 | 14
score on a scale | 17.5 (36.4) |  | 9.5 (31.6)

23. Other Pre Specified Outcome: Mood Measured by Profile of Mood States at 9 Months
Description: Profile of Mood States (POMS) is a questionnaire by MultiHealth Systems, that measures mood. In this 65 item questionnaire, subjects are asked to rate their feelings toward a statement from 0-4, with 0 being "not at all' and 4 being "extremely". There are 6 subscales which include, tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. To calculate the total mood disturbance, which is what is reported here, the subscales tension-anxiety, depression, anger-hostility, fatigue and confusion are summed and vigor is subtracted. The scale range for total mood disturbance is 200 (worst) to -32 (best). POMS will be measured after 9 months of treatment with Growth hormone in PASC subjects only.
Time Frame: 9 months
Population: mTBI and Community Control subjects complete the study at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 8.4 (29.7)

24. Other Pre Specified Outcome: Mood Measured by Profile of Mood States at 12 Months
Description: Profile of Mood States (POMS) is a questionnaire by MultiHealth Systems, that measures mood. In this 65 item questionnaire, subjects are asked to rate their feelings toward a statement from 0-4, with 0 being "not at all' and 4 being "extremely". There are 6 subscales which include, tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. To calculate the total mood disturbance, which is what is reported here, the subscales tension-anxiety, depression, anger-hostility, fatigue and confusion are summed and vigor is subtracted. The scale range for total mood disturbance is 200 (worst) to -32 (best). POMS will be measured after 9 months of treatment with Growth hormone treatment and 3 months without treatment (total 12 months) in PASC subjects only.
Time Frame: 12 months
Population: mTBI and Community Control subjects complete the study at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 14.7 (25.2)

25. Other Pre Specified Outcome: Sleep Quality Measured by Pittsburgh Sleep Quality Index at Baseline
Description: Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1 month-time interval. Minimum Score = 0 (better); Maximum Score = 21 (worse). Interpretation: Total < 5 associated with good sleep quality. Total > 5 associated with poor sleep quality. PSQI will be measured at baseline in mTBI and PASC subjects only.
Time Frame: baseline
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
score on a scale | 11.6 (4.1) |  | 9.2 (4.1)

26. Other Pre Specified Outcome: Sleep Quality Measured by Pittsburgh Sleep Quality Index at 6 Months
Description: Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1 month-time interval. Minimum Score = 0 (better); Maximum Score = 21 (worse). Interpretation: Total < 5 associated with good sleep quality. Total > 5 associated with poor sleep quality. PSQI will be measured after 6 months of treatment with growth hormone in mTBI and PASC subjects only.
Time Frame: 6 months
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 26 | 0 | 14
score on a scale | 7.5 (3.7) |  | 6.8 (4.0)

27. Other Pre Specified Outcome: Sleep Quality Measured by Pittsburgh Sleep Quality Index at 9 Months
Description: Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1 month-time interval. Minimum Score = 0 (better); Maximum Score = 21 (worse). Interpretation: Total < 5 associated with good sleep quality. Total > 5 associated with poor sleep quality. PSQI will be measured after 9 months of treatment with growth hormone in PASC subjects only.
Time Frame: 9 months
Population: mTBI and Community Control subjects complete the study at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 6.5 (2.8)

28. Other Pre Specified Outcome: Sleep Quality Measured by Pittsburgh Sleep Quality Index at 12 Months
Description: Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1 month-time interval. Minimum Score = 0 (better); Maximum Score = 21 (worse). Interpretation: Total < 5 associated with good sleep quality. Total > 5 associated with poor sleep quality. PSQI will be measured after 9 months of treatment with growth hormone and 3 months without treatment (total 12 months) in PASC subjects only.
Time Frame: 12 months
Population: mTBI and Community Control subjects complete the study at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 7.8 (4.2)

29. Other Pre Specified Outcome: Symptoms of Growth Hormone Deficiency Measured by the Questionnaire Quality of Life - Assessment of Growth Hormone Defiency in Adults at Baseline
Description: Symptoms of growth hormone deficiency will be measured in mTBI and PASC subjects using the Quality of Life - Assessment of Growth Hormone Deficiency in Adults (QoL-AGHDA). This 25-item questionnaire measures specific symptoms associated with growth hormone deficiency, with a score range of 0 to 25, with a higher score indicating worse symptoms. The QoL-ADGHA will be measured at baseline in mTBI and PASC subjects only.
Time Frame: baseline
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
score on a scale | 18.7 (4.8) |  | 15.9 (6.7)

30. Other Pre Specified Outcome: Symptoms of Growth Hormone Deficiency Measured by the Questionnaire Quality of Life - Assessment of Growth Hormone Deficiency in Adults at 6 Months
Description: Symptoms of growth hormone deficiency will be measured in mTBI and PASC subjects using the Quality of Life - Assessment of Growth Hormone Deficiency in Adults (QoL-AGHDA). This 25-item questionnaire measures specific symptoms associated with growth hormone deficiency, with a score range of 0 to 25, with a higher score indicating worse symptoms. The QoL-ADGHA will be measured after 6 months of growth hormone treatment in mTBI and PASC subjects only.
Time Frame: 6 months
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 26 | 0 | 14
score on a scale | 9.6 (8.3) |  | 11.6 (7.6)

31. Other Pre Specified Outcome: Symptoms of Growth Hormone Deficiency Measured by the Questionnaire Quality of Life - Assessment of Growth Hormone Deficiency in Adults at 9 Months
Description: Symptoms of growth hormone deficiency will be measured in PASC subjects using the Quality of Life - Assessment of Growth Hormone Deficiency in Adults (QoL-AGHDA). This 25-item questionnaire measures specific symptoms associated with growth hormone deficiency, with a score range of 0 to 25, with a higher score indicating worse symptoms. The QoL-ADGHA will be measured after 9 months of growth hormone treatment in PASC subjects only.
Time Frame: 9 months
Population: mTBI and Community Control subjects complete the study at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 8 (6)

32. Other Pre Specified Outcome: Symptoms of Growth Hormone Deficiency Measured by the Questionnaire Quality of Life - Assessment of Growth Hormone Deficiency in Adults at 12 Months
Description: Symptoms of growth hormone deficiency will be measured in PASC subjects using the Quality of Life - Assessment of Growth Hormone Deficiency in Adults (QoL-AGHDA). This 25-item questionnaire measures specific symptoms associated with growth hormone deficiency, with a score range of 0 to 25, with a higher score indicating worse symptoms. The QoL-ADGHA will be measured after 9 months of growth hormone treatment and then 3 months without treatment (total 12 months) in PASC subjects only.
Time Frame: 12 months
Population: mTBI and Community Control subjects complete the study at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 9.7 (6.2)

33. Other Pre Specified Outcome: Depression Measured by the Beck Depression Inventory-II at Baseline
Description: The Beck Depression Inventory- II assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe. The BDI will be measured at baseline in mTBI and PASC subjects only.
Time Frame: baseline
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
score on a scale | 18.9 (8.9) |  | 21.5 (11.6)

34. Other Pre Specified Outcome: Depression Measured by the Beck Depression Inventory-II at 6 Months
Description: The Beck Depression Inventory- II assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe. The BDI will be measured after 6 months of growth hormone treatment in mTBI and PASC subjects only.
Time Frame: 6 months
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 26 | 0 | 14
score on a scale | 12.1 (11.6) |  | 10.2 (10.5)

35. Other Pre Specified Outcome: Depression Measured by the Beck Depression Inventory-II at 9 Months
Description: The Beck Depression Inventory- II assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe. The BDI will be measured after 9 months of growth hormone treatment in PASC subjects only.
Time Frame: 9 months
Population: mTBI and Community Control subjects complete the study at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 8.8 (9.3)

36. Other Pre Specified Outcome: Depression Measured by the Beck Depression Inventory-II at 12 Months
Description: The Beck Depression Inventory- II assesses depressive symptom severity. The BDI-II is comprised of 21 individual items reflecting specific cognitive, affective, and physical symptoms of depression. Each item includes four statements that vary in the description of symptom of severity. Scores range from 0 to 3, with a score of "3" indicating a severe symptoms and a score of "0" indicating an absence of concern with that particular aspect of depressive symptomology. The total score is the sum of all endorsed statements. The maximum total score is 63. The BDI-II Manual designates the following raw score classifications depression severity: ≤13 = minimal; 14-19 = mild; 20-28 = moderate; ≥ 29 = severe. The BDI will be measured after 9 months of growth hormone treatment and 3 months without treatment (total 12 months) in PASC subjects only.
Time Frame: 12 months
Population: mTBI and Community Control subjects complete the study at month 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 0 | 0 | 13
score on a scale |  |  | 10.7 (8.1)

37. Other Pre Specified Outcome: Walking Distance at 25% Perceptual Effort as Measured by Walking Test at Baseline
Description: Walking performance will be assessed in mTBI and PASC patients during 6 minutes of walking in long corridor hallways. This is a standard test of walking performance that has been validated in similar studies. Here, the test will be slightly modified, with subjects asked to walk at a 25% perceived effort from minute 0 - 2, at a 50% perceived effort from minute 2 - 4, and at a 100% effort (as quickly as they can safely walk without running) from minute 4 -6. Distance traveled for each 2-minute category will be recorded. The 6-minute walking test will be completed at baseline. Measured in mTBI and PASC subjects only.
Time Frame: baseline
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
meters | 108.2 (31.3) |  | 98.3 (28.3)

38. Other Pre Specified Outcome: Walking Distance at 25% Perceptual Effort as Measured by Walking Test at 6 Months
Description: Walking performance will be assessed in mTBI and PASC patients during 6 minutes of walking in long corridor hallways. This is a standard test of walking performance that has been validated in similar studies. Here, the test will be slightly modified, with subjects asked to walk at a 25% perceived effort from minute 0 - 2, at a 50% perceived effort from minute 2 - 4, and at a 100% effort (as quickly as they can safely walk without running) from minute 4 -6. Distance traveled for each 2-minute category will be recorded. The 6-minute walking test will be completed at month 6. Measured in mTBI and PASC subjects only.
Time Frame: 6 months
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 25 | 0 | 14
meters | 118.2 (37.4) |  | 108.5 (31.7)

39. Other Pre Specified Outcome: Walking Distance at 50% Perceptual Effort as Measured by Walking Test at Baseline
Description: as for outcome 37
Time Frame: baseline
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
meters | 139.1 (30.1) |  | 125.8 (26.0)

40. Other Pre Specified Outcome: Walking Distance at 50% Perceptual Effort as Measured by Walking Test at 6 Months
Description: as for outcome 38
Time Frame: 6 months
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 25 | 0 | 14
meters | 139.3 (37.4) |  | 134.3 (28.3)

41. Other Pre Specified Outcome: Walking Distance at 100% Effort as Measured by Walking Test at Baseline
Description: as for outcome 37
Time Frame: baseline
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 28 | 0 | 17
meters | 183.6 (35.7) |  | 162.7 (24.1)

42. Other Pre Specified Outcome: Walking Distance at 100% Effort as Measured by Walking Test at 6 Months
Description: as for outcome 38
Time Frame: 6 months
Population: Community Control subjects did not complete this measure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
Number analyzed (Participants) | 25 | 0 | 14
meters | 186.6 (41.0) |  | 170.6 (27.4)

ADVERSE EVENTS:
Time Frame: mTBI arm: 6 months community control arm: 6 months PASC arm: up to 15 months
Arm/Group | mTBI Subjects | Community Control Subjects | PASC Subjects
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/27 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/27 | 0/17
Other Adverse Events (participants affected / at risk) | 26/28 | 0/27 | 17/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mTBI Subjects (N=28) | Community Control Subjects (N=27) | PASC Subjects (N=17)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 8 (8)
Hives (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Fast heartbeat (Cardiac disorders) | 5 (5) | 0 (0) | 7 (7)
Swelling (General disorders) | 16 (16) | 0 (0) | 9 (9)
Feeling Faint (Cardiac disorders) | 10 (10) | 0 (0) | 8 (8)
Injection site reactions (Skin and subcutaneous tissue disorders) | 19 (19) | 0 (0) | 8 (8)
Joint pain (Musculoskeletal and connective tissue disorders) | 20 (20) | 0 (0) | 14 (14)
Muscle soreness (Musculoskeletal and connective tissue disorders) | 19 (19) | 0 (0) | 13 (13)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 6 (6)
Pain (General disorders) | 7 (7) | 0 (0) | 3 (3)
Tingling, numbness or prickling (Nervous system disorders) | 15 (15) | 0 (0) | 12 (12)
Nausea (Gastrointestinal disorders) | 7 (7) | 0 (0) | 13 (13)
Itching (Skin and subcutaneous tissue disorders) | 7 (7) | 0 (0) | 3 (3)
Headache (General disorders) | 0 (0) | 0 (0) | 4 (4)
Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Bloating (Gastrointestinal disorders) | 5 (5) | 0 (0) | 1 (1)
Weight gain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT03554265/Prot_SAP_000.pdf